CLINICAL TRIAL: NCT04813354
Title: A Randomized, Multi-center, Open-label, Cross-over Study Comparing Critical Errors, Overall Errors, Training/Teaching Time, and Preference Attributes of the ELLIPTA Dry Powder Inhaler Versus the BREEZHALER Dry Powder Inhaler, in Adult Participants With Mild to Moderate Asthma
Brief Title: A Comparison of Critical Errors, Overall Errors, Training/Teaching Time, and Preference Attributes of the ELLIPTA Versus BREEZHALER Dry Powder Inhalers (DPIs) in Adult Participants With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 213306
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Results first posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-06

CONDITIONS: Asthma
Keywords: ELLIPTA; BREEZHALER; Dry powder inhaler; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: The study will be a randomized, multi-center, open label, placebo- controlled device handling study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ELLIPTA/ BREEZHALER/Questionnaire version 1 (Experimental): Participants received placebo ELLIPTA Dry Powder Inhaler (DPI) followed by placebo BREEZHALER DPI on Day 1. Participants were asked to complete the ease-of-use questionnaire and visual analogue scale (VAS) on their willingness to continue with the inhaler after using each device. Participants also completed the preference questionnaire version 1 on Day 1.
  Interventions: Device: ELLIPTA; Device: BREEZHALER
- ELLIPTA/ BREEZHALER/Questionnaire version 2 (Experimental): Participants received placebo ELLIPTA DPI followed by placebo BREEZHALER DPI on Day 1. Participants were asked to complete the ease-of-use questionnaire and VAS on their willingness to continue with the inhaler after using each device. Participants also completed the preference questionnaire version 2 on Day 1.
  Interventions: Device: ELLIPTA; Device: BREEZHALER
- BREEZHALER/ ELLIPTA/Questionnaire version 1 (Experimental): Participants received placebo BREEZHALER DPI followed by placebo ELLIPTA DPI on Day 1. Participants were asked to complete the ease-of-use questionnaire and VAS on their willingness to continue with the inhaler after using each device. Participants also completed the preference questionnaire version 1 on Day 1.
  Interventions: Device: ELLIPTA; Device: BREEZHALER
- BREEZHALER/ ELLIPTA/Questionnaire version 2 (Experimental): Participants received placebo BREEZHALER DPI followed by placebo ELLIPTA DPI on Day 1. Participants were asked to complete the ease-of-use questionnaire and VAS on their willingness to continue with the inhaler after using each device. Participants also completed the preference questionnaire version 2 on Day 1.
  Interventions: Device: ELLIPTA; Device: BREEZHALER

INTERVENTIONS:
Device: ELLIPTA — * ELLIPTA followed by BREEZHALER/ Preference Questionnaire version 1
  * ELLIPTA followed by BREEZHALER/ Preference Questionnaire version 2
  * BREEZHALER followed by ELLIPTA/ Preference Questionnaire version 1
  * BREEZHALER followed by ELLIPTA/ Preference Questionnaire version 2
Device: BREEZHALER — * ELLIPTA followed by BREEZHALER/ Preference Questionnaire version 1
  * ELLIPTA followed by BREEZHALER/ Preference Questionnaire version 2
  * BREEZHALER followed by ELLIPTA/ Preference Questionnaire version 1
  * BREEZHALER followed by ELLIPTA/ Preference Questionnaire version 2

SUMMARY:
This study aims to provide data in adult participants with mild to moderate asthma to assist healthcare professionals (HCPs) in assessing various attributes of ELLIPTA and BREEZHALER DPIs, by comparing the incidence of critical and overall errors, participant preference, willingness to continue with the inhaler and time to correct use. ELLIPTA® is a registered trademark of GlaxoSmithKline (GSK) and BREEZHALER® is a registered trademark of Novartis.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged 18 years or older at the time of signing the informed consent.
* Participants who have a confirmed mild or moderate asthma diagnosis as per Global Initiative for Asthma (GINA), 2020.
* Participants must be on asthma maintenance therapy (Inhaled corticosteroids [ICS] or ICS/ Long acting beta 2-agonist [LABA]) for at least 12 weeks prior to study participation.
* Participants must be naïve to both the ELLIPTA and BREEZHALER inhalers.
* Females who are not pregnant or not planning a pregnancy during the study or not Lactating.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Concurrent diagnosis of chronic obstructive pulmonary disease (COPD) or other respiratory disorders.
* History of hypersensitivity to any components of the study inhaler (e.g., lactose). In addition, participants with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates participation will also be excluded.
* Historical or current evidence of clinically significant or rapidly progressing or unstable disease that, in the opinion of the investigator, would put the safety of the participant at risk through participation, or which would affect the analysis if the disease/condition exacerbated during the study.
* Drug/alcohol abuse: Participants with a known or suspected alcohol or drug abuse, which in the opinion of the investigator could interfere with the participant's proper completion of the protocol requirement.
* A participant will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator, as well as employees of GSK or Novartis.
* Inability to Read: In the opinion of the investigator, any participant who is unable to read and/or would not be able to complete a questionnaire and understand verbal instructions.
* Medical and physical conditions that in the opinion of the investigator could impact the ability of the participant to manipulate the inhaler.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Netherlands (3):
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Nijverdal
  - GSK Investigational Site, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] van der Palen J, Slade D, Rehal S, Verma M, Plank M. A randomized, cross-over study comparing critical and overall errors, learning time, and preference of the ELLIPTA versus BREEZHALER dry powder inhalers in patients with asthma. Respir Med. 2022 Dec;205:107031. doi: 10.1016/j.rmed.2022.107031. Epub 2022 Oct 28. PMID 36368290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted across 3 centers in the Netherlands.
Pre-assignment Details: A total of 114 participants were enrolled in the study.
Period: Overall Study
Arm/Group | ELLIPTA/ BREEZHALER/Questionnaire Version 1 | ELLIPTA/ BREEZHALER/Questionnaire Version 2 | BREEZHALER/ ELLIPTA/Questionnaire Version 1 | BREEZHALER/ ELLIPTA/Questionnaire Version 2
Started | 29 | 29 | 28 | 28
Completed | 29 | 29 | 28 | 28
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ELLIPTA/ BREEZHALER/Questionnaire Version 1 | ELLIPTA/ BREEZHALER/Questionnaire Version 2 | BREEZHALER/ ELLIPTA/Questionnaire Version 1 | BREEZHALER/ ELLIPTA/Questionnaire Version 2 | Total
Number analyzed (Participants) | 29 | 29 | 28 | 28 | 114
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 1
  19-64 years | 18 | 17 | 18 | 21 | 74
  >=65 years | 10 | 12 | 10 | 7 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 12 | 15 | 17 | 65
  Male | 8 | 17 | 13 | 11 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN - SOUTH EAST ASIAN HERITAGE | 0 | 1 | 0 | 1 | 2
  WHITE - ARABIC/NORTH AFRICAN HERITAGE | 1 | 0 | 0 | 1 | 2
  WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | 28 | 28 | 28 | 25 | 109
  MIXED RACE | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Making at Least One Critical Error After Reading the Patient Information Leaflets (PIL)
Description: Participants were asked to demonstrate use of their prescribed DPI on Day 1 and any error made by the participant was recorded by the health care practitioner (HCP) in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. The errors made during demonstration by participants were defined as "critical" when an error was most likely to result in no or significantly reduced medication being inhaled. Percentage values are rounded off.
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population comprised of all participants who were randomized to study intervention in the study, completed reading of the PIL and attempted demonstration of both inhalers.
Measure: Number; unit: Percentage of participants
Groups:
- ELLIPTA DPI: Participants received placebo via the ELLIPTA DPI on Day 1 of the study. Participants were asked to complete the ease-of-use questionnaire and VAS on their willingness to continue with the inhaler after using ELLIPTA DPI. Participants also completed preference questionnaire version 1 or 2 after completing the ease-of-use questionnaire and VAS on Day 1.
- BREEZHALER DPI: Participants received placebo via the BREEZHALER DPI on Day 1 of the study. Participants were asked to complete the ease-of-use questionnaire and VAS on their willingness to continue with the inhaler after using BREEZHALER DPI. Participants also completed preference questionnaire version 1 or 2 after completing the ease-of-use questionnaire and VAS on Day 1.
Arm/Group | ELLIPTA DPI | BREEZHALER DPI
Number analyzed (Participants) | 114 | 114
Percentage of participants | 6 | 26
Statistical Analysis 1: Comparison: ELLIPTA DPI vs BREEZHALER DPI; Test type: Superiority; p < 0.001, Exact conditional logistic regression; Odds Ratio (OR) = 0.11, 95% CI 2-sided [0.01 to 0.40] — Odds ratio between ELLIPTA DPI and BREEZHALER DPI was calculated using an exact conditional logistic regression model with participant as fixed strata, inhaler and period as fixed effects

2. Secondary Outcome: Percentage of Participants Making at Least One Critical Error After Receiving Further Instructions (up to 3) From HCP
Description: Participants were asked to demonstrate inhaler use after reading PIL. The errors made during demonstration by participants were defined as "critical" when an error was most likely to result in no or significantly reduced medication being inhaled. If the participant made any error according to the error checklists, the HCP provided instructions on the correct use of the inhaler to the participant and the participant was then asked to demonstrate the inhaler use again. Any error made by the participant were recorded by the HCP in the checklist. The same procedure was repeated if the participant continued to make errors in the use of the inhaler. In total, the HCP provided up to 3 instructions on the use of the inhaler. Same procedure was followed for second inhaler. Percentage of participants making at least one critical error after receiving 1st instruction, 2nd instruction and 3rd instruction from HCP were reported. Percentage values are rounded off.
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population
Measure: Number; unit: Percentage of participants
Arm/Group | ELLIPTA DPI | BREEZHALER DPI
Number analyzed (Participants) | 114 | 114
Percentage of participants
  After 1st Instruction by HCP | 1 | 4
  After 2nd Instruction by HCP | 0 | 0
  After 3rd Instruction by HCP | 0 | 0

3. Secondary Outcome: Percentage of Participants Making at Least One Overall Error After Reading PIL
Description: Participants were asked to demonstrate use of their prescribed DPI on Day 1 and any error made by the participant was recorded by the HCP in the checklist. Checklist of instructions for correct use were based on the steps for correct use listed in PILs for the respective DPI. An overall error was any error in inhaler technique which includes a critical and non-critical error. Percentage values are rounded off.
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population
Measure: Number; unit: Percentage of participants
Arm/Group | ELLIPTA DPI | BREEZHALER DPI
Number analyzed (Participants) | 114 | 114
Percentage of participants | 27 | 41
Statistical Analysis 1: Comparison: ELLIPTA DPI vs BREEZHALER DPI; Test type: Other; p = 0.005, Exact conditional logistic regression; Odds Ratio (OR) = 0.25, 95% CI 2-sided [0.03 to 0.74] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants Making at Least One Overall Error After Receiving Further Instructions (up to 3) From the HCP
Description: Participants were asked to demonstrate inhaler use after reading PIL. If the participant made any error according to the error checklists, the HCP provided instructions on the correct use of the inhaler to the participant and the participant was then asked to demonstrate the inhaler use again. Any error made by the participant were recorded by the HCP in the checklist. The same procedure was repeated if the participant continued to make errors in the use of the inhaler. In total, the HCP provided up to 3 instructions on the use of the inhaler. Same procedure was followed for second inhaler. An overall error was any error in inhaler technique which includes a critical and non-critical error. Percentage of participants making at least one overall error after receiving 1st instruction, 2nd instruction and 3rd instruction from HCP were reported. Percentage values are rounded off.
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population
Measure: Number; unit: Percentage of participants
Arm/Group | ELLIPTA DPI | BREEZHALER DPI
Number analyzed (Participants) | 114 | 114
Percentage of participants
  After 1st Instruction by HCP | 3 | 9
  After 2nd Instruction by HCP | 0 | 1
  After 3rd Instruction by HCP | 0 | 0

5. Secondary Outcome: Number of Critical and Overall Errors Made by Participants After Reading PIL and After Receiving Further Instructions (up to 3) From HCP
Description: Participants were asked to demonstrate inhaler use after reading PIL. If participant made any error according to error checklists, the HCP provided instructions on correct use of inhaler to participant and participant was then asked to demonstrate inhaler use again. Critical error was any error which most likely to result in no or significantly reduced medication being inhaled. An overall error was any error in inhaler technique, which includes a critical and non-critical. Any error made by the participant was recorded by the HCP in checklist. The same procedure was repeated if the participant continued to make errors in the use of inhaler. In total, HCP provided up to 3 time instructions on correct use of inhaler. Same procedure was followed for second inhaler. The number of critical and overall errors made by participants after reading PIL and after receiving 1st instruction, 2nd instruction and 3rd instruction from HCP were reported.
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population
Measure: Number; unit: Errors
Arm/Group | ELLIPTA DPI | BREEZHALER DPI
Number analyzed (Participants) | 114 | 114
Errors
  Critical Errors; After reading PIL | 7 | 47
  Critical Errors; After 1st instruction | 1 | 8
  Critical Errors; After 2nd instruction | 0 | 0
  Critical Errors; After 3rd instruction | 0 | 0
  Overall Errors; After reading PIL | 44 | 121
  Overall Errors; After 1st instruction | 3 | 18
  Overall Errors; After 2nd instruction | 0 | 3
  Overall Errors; After 3rd instruction | 0 | 0

6. Secondary Outcome: Percentage of Participants Who Required Further Instruction (up to 3) From HCP to Demonstrate Correct Inhaler Use
Description: Participants were asked to demonstrate inhaler use after reading PIL. If the participant made any error according to the error checklists, the HCP provided instructions on the correct use of the inhaler to the participant and the participant was then asked to demonstrate the inhaler use again. Any error made by the participant were recorded by the HCP in the checklist. The same procedure was repeated if the participant continued to make errors in the use of the inhaler. In total, the HCP provided up to 3 times instructions on the correct use of inhaler. Same procedure was followed for second inhaler. Percentage of participants who required zero, 1st, 2nd and 3rd instruction from HCP to demonstrate correct inhaler use were reported. Percentage values are rounded off.
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population
Measure: Number; unit: Percentage of participants
Arm/Group | ELLIPTA DPI | BREEZHALER DPI
Number analyzed (Participants) | 114 | 114
Percentage of participants
  Zero instructions | 73 | 59
  1st instruction | 25 | 32
  2nd instruction | 3 | 8
  3rd instruction | 0 | 1

7. Secondary Outcome: Time Taken to Demonstrate Inhaler Use After Reading PIL Without HCP Intervention (T1)
Description: Participants were asked to demonstrate inhaler use after reading PIL and any error made by the participant was recorded by the HCP in the checklist. Time taken to demonstrate inhaler use after reading PIL without HCP intervention was the amount of time taken to correctly demonstrate inhaler use without HCP intervention. T1 was calculated from the start of inhaler demonstration by the participant after reading the PIL until completion of the first attempt.
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population. Only those participants with data available at specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | ELLIPTA DPI | BREEZHALER DPI
Number analyzed (Participants) | 83 | 67
Minutes | 1.00 [0.00 to 2.00] | 2.00 [2.00 to 4.00]

8. Secondary Outcome: Time Taken to Give Instructions by HCP on the Use of Inhaler and to Demonstrate the Correct Inhaler Use (T2)
Description: Time taken by HCP to demonstrate the correct use of inhaler was the time from when the HCP started to instruct the participant until correct use was demonstrated. It includes the time used by the HCP for re-instructing the participants throughout. T2 was calculated from the first instruction provided by the HCP until demonstration of correct use. Up to 3 further attempts were made after completion of the first attempt.
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | ELLIPTA DPI | BREEZHALER DPI
Number analyzed (Participants) | 114 | 114
Minutes | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 2.00]

9. Secondary Outcome: Total Time Taken for Demonstration of Correct Use After Reading PIL (T1+T2)
Description: Participants were asked to demonstrate inhaler use after reading PIL and any error made by the participant was recorded by the HCP in the checklist. Total time taken for demonstration of correct use after reading PIL was the time from when the participant started the demonstration until correct use is demonstrated (4 attempts= once after the reading the PIL and following instruction from investigator up to 3 times). T1+T2 was calculated from the start of inhaler demonstration after reading the PIL until correct demonstration was observed.
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | ELLIPTA DPI | BREEZHALER DPI
Number analyzed (Participants) | 114 | 114
Minutes | 1.00 [0.00 to 1.00] | 2.00 [2.00 to 4.00]

10. Secondary Outcome: Number of Participants Assessed for Ease-of-use of ELLIPTA Inhaler and BREEZHALER Inhaler Using Questionnaire (Grouped as 'Very Easy', 'Easy', 'Neutral', 'Difficult' and 'Very Difficult')
Description: Participant were asked to complete the ease of use questionnaire for the DPI once error assessment of each inhaler was completed. This was a series of 6 questions (Ease of use rating, Telling how many doses were left in inhaler, Learning how to use inhaler, Handling the inhaler, Preparing inhaler and Holding inhaler while using it). Each question had one response to choose from 5 options of ease of use (Very easy, easy, neutral, difficult and very difficult). Participants were asked to rate based on their ease of use experience with device using a scale ranging from 1 (very easy) to 5 (very difficult). A higher rating indicated that the inhaler was difficult to use and a lower rating indicated that inhaler was easier to use. This questionnaire was completed for the first device before moving to the critical errors assessment of the second device. Data has been categorized and reported as 'Very easy', 'Easy', 'Neutral', 'Difficult' and 'Very Difficult' with respect to each question.
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | ELLIPTA DPI | BREEZHALER DPI
Number analyzed (Participants) | 114 | 114
Participants
  Ease of use of inhaler, Very Easy | 64 | 18
  Ease of use of inhaler, Easy | 43 | 41
  Ease of use of inhaler, Neutral | 5 | 28
  Ease of use of inhaler, Difficult | 2 | 26
  Ease of use of inhaler, Very difficult | 0 | 1
  Ease of telling number of doses left, Very easy | 85 | 35
  Ease of telling number of doses left, Easy | 27 | 47
  Ease of telling number of doses left, Neutral | 2 | 19
  Ease of telling number of doses left, Difficult | 0 | 11
  Ease of telling number of dose left,Very difficult | 0 | 2
  Ease of learning how to use inhaler, Very easy | 63 | 28
  Ease of learning how to use inhaler, Easy | 47 | 41
  Ease of learning how to use inhaler, Neutral | 2 | 27
  Ease of learning how to use inhaler, Difficult | 2 | 17
  Ease of learning how to use inhaler,Very difficult | 0 | 1
  Ease of handling the inhaler, Very easy | 67 | 24
  Ease of handling the inhaler, Easy | 42 | 44
  Ease of handling the inhaler, Neutral | 3 | 28
  Ease of handling the inhaler, Difficult | 2 | 17
  Ease of handling the inhaler, Very difficult | 0 | 1
  Ease of preparing the inhaler for use,Very easy | 70 | 19
  Ease of preparing the inhaler for use, Easy | 42 | 45
  Ease of preparing the inhaler for use, Neutral | 2 | 26
  Ease of preparing the inhaler for use, Difficult | 0 | 21
  Ease of preparing the inhaler for use, Very difficult | 0 | 3
  Ease of holding inhaler while using, Very easy | 56 | 31
  Ease of holding inhaler while using, Easy | 47 | 53
  Ease of holding inhaler while using, Neutral | 7 | 21
  Ease of holding inhaler while using, Difficult | 3 | 9
  Ease of holding inhaler while using,Very difficult | 1 | 0

11. Secondary Outcome: Number of Participants Assessed for Ease-of-use of ELLIPTA Inhaler and BREEZHALER Inhaler Using Questionnaire (Grouped as 'Easy' and 'Difficult')
Description: The ease-of-use questionnaire consists of a series of 6 questions (Ease of use rating, Telling how many doses were left in inhaler, Learning how to use inhaler, Handling inhaler, Preparing inhaler and Holding inhaler while using it). Each question had one response to choose from 5 options of ease of use(Very easy, easy, neutral, difficult and very difficult). Participants were asked to rate based on their ease of use experience with device using a scale ranging from 1(very easy) to 5(very difficult). A higher rating indicated that inhaler was difficult to use and a lower rating indicated that inhaler was easy to use. This questionnaire was completed for first device before moving to critical errors assessment of second device. Participant who responded Very Easy or Easy was considered Easy and participant who responded Neutral, Difficult or Very Difficult was considered Difficult. Data has been categorized and reported as Easy and Difficult with respect to each question
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | ELLIPTA DPI | BREEZHALER DPI
Number analyzed (Participants) | 114 | 114
Participants
  Ease of use of inhaler, Easy | 107 | 59
  Ease of use of inhaler, Difficult | 7 | 55
  Ease of telling number of doses left,Easy | 112 | 82
  Ease of telling number of doses left, Difficult | 2 | 32
  Ease of learning how to use inhaler, Easy | 110 | 69
  Ease of learning how to use inhaler, Difficult | 4 | 45
  Ease of handling the inhaler, Easy | 109 | 68
  Ease of handling the inhaler, Difficult | 5 | 46
  Ease of preparing the inhaler for use, Easy | 112 | 64
  Ease of preparing the inhaler for use, Difficult | 2 | 50
  Ease of holding inhaler while using it, Easy | 103 | 84
  Ease of holding inhaler while using it, Difficult | 11 | 30

12. Secondary Outcome: Visual Analogue Scale (VAS) for the Assessment of Participants Willingness to Continue With the Inhaler
Description: Participants were asked the question regarding their willingness to continue with the inhaler using a visual analogue scale ranging from 0 (not willing) to 100 (definitely willing) after completion of the critical errors assessment for each inhaler and the ease of use questionnaire for that inhaler. Participants marked on the VAS scale, how willing they were to continue using the inhaler. That mark was measured with a ruler to determine the numerical score. It ranges from 0 to 100 where, higher score on the scale indicates better outcome, means participant was definitely willing to continue using the inhaler.
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | ELLIPTA DPI | BREEZHALER DPI
Number analyzed (Participants) | 114 | 114
Scores on a scale | 79.9 (24.30) | 52.3 (30.86)
Statistical Analysis 1: Comparison: ELLIPTA DPI vs BREEZHALER DPI; Test type: Other; p < 0.001, Paired samples t-test; Mean Difference (Final Values) = 27.63, 95% CI 2-sided [21.31 to 33.96]

13. Secondary Outcome: Number of Participants With Inhaler Preferences Assessed Using Preference Questionnaire
Description: Participants were asked to complete the assigned preference questionnaires after completing the errors in use assessment for both devices. Participants were asked to provide their responses in terms of their preference to the ELLIPTA inhaler or BREEZHALER inhaler or No preference. Participants preference was assessed using series of 7 questions (Preferred inhaler-overall, Preference based on the number of steps to take the medication, Preference based on the time needed to take the medication, Preference based on how easy the inhaler was to use, Preference based on the size of the inhaler, Preference based on the comfort of the mouthpiece and Preference based on the ease of opening the inhaler). Participants had to choose one response from 3 preference options (ELLIPTA inhaler or BREEZHALER inhaler or No preference).
Time Frame: Day 1
Population: Modified intention-to-treat (mITT) Population. Data has been presented for All treated participants in a single arm as the intent of this endpoint was to assess the participant's preference to the inhaler (among both the inhalers) that was used.
Measure: Count of Participants; unit: Participants
Groups:
- All Treated Participants: Participants received placebo via the ELLIPTA DPI and via BREEZHALER DPI on Day 1. Participants were asked to complete the ease-of-use questionnaire and VAS on their willingness to continue with the inhaler after using each device. Participants also completed preference questionnaire versions 1 or 2 after completing the ease-of-use questionnaire and VAS.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 114
Participants
  Preferred inhaler- overall; ELLIPTA | 85
  Preferred inhaler- overall;BREEZHALER | 19
  Preferred inhaler- overall;No preference | 10
  Preference by Number of Steps Needed;ELLIPTA | 99
  Preference by Number of Steps Needed;BREEZHALER | 5
  Preference by Number of Steps Needed;No preference | 10
  Preference based on time needed,ELLIPTA | 90
  Preference based on time needed,BREEZHALER | 6
  Preference based on time needed;No preference | 18
  Preference based on How Easy to Use;ELLIPTA | 94
  Preference based on How Easy to Use;BREEZHALER | 11
  Preference based on How Easy to Use;No preference | 9
  Preference based on Size;ELLIPTA | 58
  Preference based on Size;BREEZHALER | 39
  Preference based on Size;No preference | 17
  Preference based on Comfort;ELLIPTA | 52
  Preference based on Comfort;BREEZHALER | 41
  Preference based on Comfort;No preference | 21
  Preference based on Ease of Opening;ELLIPTA | 80
  Preference based on Ease of Opening;BREEZHALER | 13
  Preference based on Ease of Opening;No preference | 21

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-serious AEs (non-SAEs) were collected on Day 1 of the study
Description: Full Analysis Set Population was used to assess All-cause mortality, SAEs and non-SAEs, which comprised of all randomized participants who used at least one study inhaler.
Arm/Group | ELLIPTA DPI | Breezhaler DPI
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/114
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/114
Other Adverse Events (participants affected / at risk) | 0/114 | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT04813354/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT04813354/SAP_001.pdf